CLINICAL TRIAL: NCT07237490
Title: In Our Prospective and Randomized Controlled Study, 42 Children With Unilateral Cerebral Palsy Were Included and Randomized as the mCIMT Group Delivered Via Telerehabilitation (n=21) and the Control Group (n=21). The First Group Received mCIMT Treatment Together With Telerehabilitation for 1 Hour, 3 Times a Week for 6 Weeks. In Addition, 30 Minutes of Indoor Activity Practices Were Performed Every Day. The Second Group Received a Home Program Under the Supervision of Parents for 1 Hour, 3 Times a Week for 6 Weeks.
Brief Title: Effectiveness of Modified Constraint-Induced Movement Therapy Delivered Via Telerehabilitation in Children With Unilateral Cerebral Palsy: A Prospective Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Mustafa Hakan KAPUCU, Medical Doctor (Res. Assist. Dr.), Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2480576
Record Dates: First submitted 2025-09-24; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-07

CONDITIONS: mCIMT Effect Via Telerehabilitation
Keywords: Cerebral palsy, telerehabilitation , mCIMT, exercise, hand functions
MeSH Terms: conditions — Cerebral Palsy; Motor Activity

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Controlled Trial - Single Blinded
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- via Telerehabilitation mCIMT (Active Comparator): The first group received mCIMT treatment together with Telerehabilitation for 1 hour, 3 times a week for 6 weeks. In addition, 30 minutes of indoor activity practices were performed every day.
  The second group received a home program under the supervision of parents for 1 hour, 3 times a week for 6 weeks.
  Interventions: Other: mCIMT via Telerehabilitation
- home exercises control group (Active Comparator): A 1-hour home program will be implemented 3 days a week.
  Interventions: Other: home exercise program

INTERVENTIONS:
Other: mCIMT via Telerehabilitation — In this group, patients aged 4-12 with unilateral cerebral palsy received mCIMT via the Eczacıbaşı EVITAL app for upper extremity rehabilitation. For six weeks, they performed mCIMT three times a week for one hour under therapist supervision and with parental supervision, two times a week for one hour under parental supervision, and half an hour each day of selected daily activities using the affected extremity, with gloves on the unaffected extremity.
  Arms: via Telerehabilitation mCIMT
Other: home exercise program — Patients in this group with unilateral CP underwent a home exercise program, which they continued for one hour, three days a week.
  The upper extremity exercise program included range of motion exercises, stretching exercises, activities of daily living exercises, and play-based exercises.
  This program lasted an average of 60 minutes.
  Arms: home exercises control group

SUMMARY:
Aim:In this prospective and randomized controlled thesis study; we aimed to compare Modified Constraint-Induced Movement Therapy (mCIMT) delivered via Telerehabilitation with the home program in children with Unilateral Cerebral Palsy (CP) and to determine whether Telerehabilitation has a positive effect on upper extremity functions and quality of life.

Method: In our prospective and randomized controlled study, 42 children with unilateral cerebral palsy were included and randomized as the mCIMT group delivered via Telerehabilitation (n=21) and the control group (n=21).

The first group received mCIMT treatment together with Telerehabilitation for 1 hour, 3 times a week for 6 weeks. In addition, 30 minutes of indoor activity practices were performed every day.

The second group received a home program under the supervision of parents for 1 hour, 3 times a week for 6 weeks.

.In the randomized double-blind study, initial assessments, post-treatment and follow-up assessments were performed by the researcher who was blinded to the group distribution.

The primary outcome measure was the Assisting Hand Assessment (AHA), which was used to evaluate upper extremity function. The researcher administering this assessment was blinded to group allocation. Secondary outcome measures included the Modified Jebsen Taylor Hand Function Test, range of motion assessed with a goniometer, spasticity evaluated using the Modified Ashworth Scale, grip strength measured with a Jamar dynamometer, manual ability classified using the Manual Ability Classification System (MACS), activities of daily living assessed by ABILHAND-Kids, and quality of life evaluated using the KINDL questionnaire.

Post-treatment assessments were performed at the beginning of the study and 6 weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion between the ages of 4-12
* Diagnosis of unilateral CP by a specialist
* Ability to extend the suspected wrist more than 10°
* Demonstration of ability to follow simple commands and participation in assigned tasks
* Gross Motor Function Classification System Level 1 or 2
* Manual Skills Classification System Level 1, 2 or 3
* Muscle tone is normal/mild/moderate (Modified Ashworth Scale level 0-1-2)
* No contractures in the upper extremity
* Agrees to attend intensive therapy sessions and to stop all other upper extremity therapeutic interventions for the 3-month follow-up period

Exclusion Criteria:

* Significant contractures in the wrist, elbow, and fingers that prevent daily activities
* Lack of active movement in the affected upper extremity
* Cognitive impairment that causes inability to understand and perform simple commands and tasks
* Inability to continue treatment protocol due to school schedule
* Uncontrolled disease (endocrinologic, cardiovascular, pulmonary, hematologic, hepatic, renal), active systemic inflammatory disease, and/or history of malignancy
* Current or previous treatments not compatible with the study treatment protocol
* Orthopedic surgery (tendon transfer/tendon lengthening) performed on the affected upper extremity
* Botulinum toxin injection into upper extremity muscles within the last 6 months
* Dorsal rhizotomy
* Intrathecal baclofen pump

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2023-12-12 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-09-25 (Actual)

PRIMARY OUTCOMES:
Assisting Hand Assessment | before treatment and 6 weeks after treatment
  The AHA is a test that measures how patients with upper extremity dysfunction, such as hemiplegic CP or congenital brachial plexus injury, use their affected hand in conjunction with their unaffected hand during two-handed play. It was first validated in children aged 18 months to 5 years (Small Kids AHA), and then two play tables were created for children aged 6 to 12 years (School Kids AHA). In this assessment method, a camera records the child performing tasks and playing with both hands. This assessment method can be administered by healthcare professionals who have completed the training and received certification. The test consists of two stages: first, the assessor (therapist, physician) sits opposite the child, and an environment is prepared using age-appropriate toys from the AHA kit to enable the child to perform all upper extremity functions using both hands. A camera positioned behind the assessor records this process.

SECONDARY OUTCOMES:
ABILHAND KIDS | before treatment and 6 weeks after treatment
  ABILHAND-Kids is a scale that assesses the extent to which children with cerebral palsy can use their manual skills in daily living activities such as self-care, and the difficulties perceived by parents during these activities.
Modified Jebsen-Taylor Hand Function Test | before treatment and 6 weeks after treatment
  The Jebsen-Taylor Hand Function Test (JFTT) is a standardized performance test developed to assess unimanual daily skills. In this test, children are asked to perform tasks such as grasping, releasing, and moving objects at varying levels of difficulty as quickly and accurately as possible. The assessment time is recorded in seconds.
Joint Range of Motion | before treatment and 6 weeks after treatment
  In our study, ROM in the affected extremity was measured separately using a joint goniometer, both actively and passively, for finger flexion/extension, wrist flexion/extension, supination/pronation, elbow flexion/extension, and shoulder flexion/extension/abduction/adduction/internal rotation/external rotation.
Grip Strength | before treatment and 6 weeks after treatment
  Grip strength was measured separately in both upper extremities using a Baseline® Smedley spring dynamometer (child, 110 lb, USA).
  The standard procedure outlined by Mathiowetz et al. was followed during the assessment: three maximum voluntary grips were performed for each hand. The average of these three measurements was taken, and the results were recorded in kilograms of force (kgF).
Modified Ashworth Scale | before treatment and 6 weeks after treatment
  Muscle tone was assessed in five major muscle groups in the affected upper extremity. The Modified Ashworth Scale (MAS) was used, and muscle tone was graded from 0 (normal) to 4 (significantly increased).
  The muscle groups assessed were: elbow flexors, elbow extensors, wrist flexors, wrist extensors, and finger flexors.
KINDL | before treatment and 6 weeks after treatment
  The Children's General Health-Related Quality of Life Scale (KINDL-R) is a self-report scale developed to assess the health-related quality of life of children and adolescents. It is available in three versions to suit different age groups: the Kiddy-KINDL-R (interviewer-administered version) for children aged 4-7, the Kid-KINDL-R for children aged 8-12, and the Kiddo-KINDL-R for adolescents aged 13-16. In addition, two parent forms are available that allow families to indirectly assess the quality of life of younger children (ages 4-7) and older children and adolescents (ages 8-16).

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe R AYDIN, Professor Doctor, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided